CLINICAL TRIAL: NCT06057883
Title: Effects of Probiotics Formulation on Stress and Skin Health in Younger Adult Females: A Holistic Approach to Skin Health, an Open-Label Proof-of-Concept Study
Brief Title: Effects Of A Probiotic Formulation On Stress and Skin Health in Younger Adult Females
Acronym: Cosmebiome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: Laboratoire Cosderma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: L-028
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stress; Skin Imperfections; Skin Fine Lines
Keywords: Psychobiotic; Probiotics; Perceived Stress; Young Females; Skin; Fine Lines; Hydration; Firmness; Skin Tone; Holistic
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A Single Arm, Open-Label, and Proof-of-Concept Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic arm (Experimental): All participants will be given the active probiotic product as this is a single arm, open-label study.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — A blend of two probiotic strains. Participants will take 1 capsule daily at 3 billion Colony Forming Units (CFUs)

SUMMARY:
The goal of this clinical trial is to test to efficacy of a probiotic blend on stress and skin appearance in young females. It is hypothesized that those taking the probiotic blend will have decreased levels of perceived stress and this will be reflected positively on their skin appearance.

DETAILED DESCRIPTION:
The goal of this open-label clinical trial is to evaluate the potential beneficial effects of a probiotic formulation on mental wellbeing and skin appearance in healthy young adult females in line with the holistic approach context and beauty from within principle. The main questions it aims to answer are related to:

* Probiotics effects on stress.
* Probiotics effects on sleep quality.
* Probiotics effects on skin appearance (fine lines and skin tone) and parameters (hydration and firmness) Participants will be recruited and, if consenting and eligible, will be provided with the probiotic capsules and instructed to ingest one capsule daily, preferably in the evening for 56 consecutive days. In-person visits will take place at baseline, mid-intervention (Day 28), and end of intervention (Day 56) to carry out assessment activities at Cosderma site.

Researchers will compare the outcome assessment measures after the probiotic ingestion to baseline values to highlight any significant effects or trends.

ELIGIBILITY:
Inclusion Criteria:

Each participant must fulfill all the inclusion criteria below:

1. Females between 30 to 45 years old, inclusive.
2. Caucasian type.
3. Normal to dry skin to the face (excluded very dry skin).
4. Have a regular menstrual cycle (participants not known to have hormonal imbalance, be in the pre-menopausal or menopausal state).
5. Have a skin phototype I, II or III.
6. Have a negative urine pregnancy test at screening and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months, and participants must agree to sign a release form (Appendix 4).

   Other acceptable methods of birth control include:
   * Abstinence or agrees to use contraception if planning to become sexually active
   * Hormonal contraceptives
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle
   * Vasectomy of partner at least 6 months prior to screening
7. Able to give free, informed and express consent to participate,
8. Affiliated with social security in accordance with the recommendations of the French law (Loi Jardé: n° 2016-1537 - 16.11.16) concerning biomedical research.
9. Visible fine to moderate fine lines on at least one area of the face (e.g., forehead, or crow's feet area, etc.) as assessed by a score ≥ 2 and ≤ 6 on a 10-point clinical scale.
10. Corneometer® on the face as assessed by an index > 20 and ≤ 60.
11. Corneometer® on the forearms as assessed by an index ≤ 50.
12. 50% of the participants fulfilling all inclusion criteria and, in addition, self-reported having a sensitive skin.
13. Does not plan to expose face to sunlight during the study.
14. Willingness to maintain eating habits for the duration of the study (quick check of diet: sugar/protein/fat/fruit intake and average drink consumption).
15. Willing to refrain from using any cream and/or makeup on the face, eyes, lips, or palms for study visits and photo capture.
16. Participants are otherwise healthy and in a good general health and mental health.
17. Willing to discontinue consumption of probiotic supplements, probiotic fortified products, and fiber supplements for the duration of the study.
18. Willingness to maintain the same skin care routine for the duration of the study.
19. Willingness to complete all study visits, assessment questionnaires, and diaries.

Exclusion Criteria:

Eligible participants must not meet any of the non-inclusion criteria below:

1. Currently pregnant, or breast feeding, or planning to be pregnant during the study.
2. Current smoker.
3. Suffering from a chronic or acute skin condition on the face and forearms (atopic dermatitis, acne, eczema, psoriasis, rash, severe dryness, etc.), unless the condition is deemed stabilized and will not affect study outcomes or be negatively affected by the intervention in the opinion of the investigator.
4. Current use of antiaging products, unless the participant has been using the same product, with the same frequency and concentration for the past ≥ 3 months.
5. Introduction of a new antiaging product during the study, or a change in the frequency or concentration of a routinely used antiaging product.
6. Introduction of new skin care products during the study, unless medically prescribed.
7. Facial surgery 5 years before study start.
8. Chemical treatment (e.g., Botox injection) within 1 year before study start.
9. Frequent UV exposure or expect high exposure to the sun during the study.
10. Diagnosed with a general physical or mental health problem (e.g., diabetes, peptic ulcer, inflammatory bowel disease, depression, anxiety, insomnia, etc.) or systemic disease that may pose a safety risk, interfere with the dietary intake of the investigational product, or impact the assessment of study outcomes.
11. Diagnosed with an autoimmune disease or are immune compromised due to medical condition or medications intake (e.g., acquired immunodeficiency (HIV), organ transplant, lymphoma, chemotherapy, chronic corticosteroids intake, etc.).
12. Currently taking oral or local anti-inflammatory treatment or have been taken daily anti-inflammatory therapy in the 2 weeks preceding the inclusion visit. Note: participants could be eligible to participate after a 2-week washout period.
13. Currently on corticosteroid treatment or antihistamines or other dermatological treatment or specialties based on vitamin A acid or its derivatives in the 2 weeks preceding the study. Note: participants could be eligible to participate after a 2-week washout period.
14. Treated with an oral retinoid within 6 months prior to the study.
15. Subjects who have applied make-up products to the face and forearms the day of the inclusion visit.
16. Subjects who have washed their face and forearms with any other means than clear water (no soap or cleanser) on the day of the inclusion visit.
17. Applied self-tanning products to the face and forearms within 2 weeks preceding the inclusion visit. Note: participants could be eligible to participate after a 2-week washout period.
18. Have eyelashes extensions.
19. Applied a moisturizing product (hygiene moisturizing product or care product) on the face and forearms within the last 48 hours.
20. Wearing tight clothing that do not let the forearms show.
21. Performed hair removal on the forearms within the last 48 hours.
22. Have cutaneous marks on the face and forearms which could interfere with the skin's clinical signs assessment (pigmentation issues, scar tissues, over-developed hairiness, too many ephelides and naevi, sunburns, tattoos, etc.).
23. Currently using a supplement that could affect study outcomes such as melatonin.
24. Use of probiotics other than the study supplement within 1 month of the inclusion visit. Note: participants could be eligible to participate after a 4-week washout period.
25. Use of any antibiotic drug within 1 month of the inclusion visit. Note: participants could be eligible to participate after a 4-week washout period.
26. Subjects working as staff at Cosderma.
27. Intending to be vaccinated during the study period.
28. Currently enrolled or intending to be enrolled in another trial during the study period, or not meeting their 2 weeks exclusion period since their last participation in a study.
29. Subjects who have been deprived of their liberty by administrative or legal decision or under judicial supervision.
30. Subjects who could not be contacted in an emergency by phone.
31. Milk or soy allergy or severe lactose intolerance.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
The effect of the probiotic intake on perceived stress levels. | 56 Days
  The change from baseline in the level of perceived stress will be assessed by the 10-item perceived stress scale (PSS-10) questionnaire before consumption of the probiotic (baseline) then after 28 and 56 days of intake.
  The PSS-10 is a widely used self-report questionnaire that measures the degrees to which individuals perceive their lives as unpredictable, uncontrollable, and overloaded. The scale consists of 10 items, which assess the individual's feelings and thoughts related to stress in the past month. The items are designed to capture both positive and negative aspects of stress, including factors such as feeling nervous or stressed, feeling confident in handling personal problems, and feeling that things are going well. The PSS-10 has been extensively used in research studies and clinical settings and has been found to have good reliability and validity.

SECONDARY OUTCOMES:
The effect of the probiotic intake on sleep quality. | 56 Days
  Participants will be asked to complete the 3-item questionnaire adapted from the Canadian Health Measures Survey before consumption of the probiotic (baseline) then after 28 and 56 days of intake.
  This is not a validated questionnaire; the questions were administered to assess subjective sleep quality among Canadians by Statistics Canada.
  For each item, the percentage of each answer will be calculated and compared to baseline at Day 28 (mid-intervention) and Day 56 (end of intervention).
The effect of the probiotic intake on skin hydration. | 56 Days
  The hydration level of the upper layers of the epidermis will be assessed with the Corneometer CM825® which runs at frequencies between 0.9 and 1.2 MHz. Corneometric index (M) will be reported in units ranging from 5 to 125. The moisturizing effect will be evaluated by comparing measurements taken at baseline and after intervention (at 28 and 56 Days).
The effect of the probiotic intake on skin firmness. | 56 Days.
  Skin firmness will be assessed by Cutometer®. The device generates a negative pressure which can vary between 20 up to 500 mbar.
  The skin is sucked up inside the probe for 2 seconds with a constant negative pressure.Then the pressure stops, and the skin returns to its initial state. Values obtained at Day 28 and Day 56 twill be compared to baseline.
The effect of the probiotic intake on facial fine lines appearance. | 56 Days
  Facial fine lines will be clinically assessed by an experienced technician on a 10-point scale. Assessment will take place on the whole face, forehead, and crow's feet area (0 = no visible fine lines, 9 = very visible fine lines). Assessment will take place at Evalux bench® (Orion concept) with the 3 neon lights (2 lateral and 1 horizontal) turned on.
  Score recorded at Day 28 and 56 will be compared to baseline.
The effect of the probiotic intake on skin tone appearance. | 56 Days
  Facial skin tone will be clinically assessed by an experienced technician on a 10-point scale. Assessment will take place on uniformity (0 = Non-uniform complexion, 9 = Very uniform complexion), and radiance (0 = Non-glowy complexion , 9 = Glowy complexion).
  Assessment will take place at Evalux bench® (Orion concept) with the 3 neon lights (2 lateral and 1 horizontal) turned on, except for the radiance assessment which will take place without the neon lights and only with the light of the room.
  Score recorded at Day 28 and 56 will be compared to baseline.
The effect of the probiotic intake on general skin appearance. | 56 Days
  Photographs of the front face and one profile will be taken by Visia-CR® camera. Images will be taken at two settings standard and polarized light.
  All images will be sent to the Sponsor. No statistical analysis will be performed. Picture will be used for illustrative purpose only.
Overall participants' satisfaction with the intervention. | 56 Days
  Participants will be asked to complete a self-administered questionnaire designed to assess participant's satisfaction with the product after 28 and 56 days of intake.
  This questionnaire is written by Cosderma in collaboration with the Sponsor. The answering modalities will be the following: "strongly agree", "somewhat agree", "somewhat disagree", "strongly disagree". A "Non-applicable" option will be added when needed.
The effect of the probiotic intake on Gastro-Intestinal (GI) health. | 56 Days.
  Participants will be asked to complete the 15-item gastrointestinal symptom rating scale (GSRS) questionnaire before starting intervention (baseline) then after 28 and 56 days of intervention.
  GSRS is a widely used and validated tool. This self-administered questionnaire is designed to assess the frequency and severity of gastrointestinal (GI) symptoms. It consists of 15 items, which are grouped into five subscales:
  1. Abdominal pain
  2. Reflux syndrome
  3. Indigestion syndrome
  4. Diarrhea syndrome
  5. Constipation syndrome Average total scores at Day 28 (mid-intervention) and Day 56 (end of intervention) will be compared to baseline.
The probiotic's safety and tolerability. | 56 Days
  Incidence of clinical events (sensations of discomfort or clinical signs) occurring during the study after the consumption of the probiotic.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Milpied, Principal Investigator — Laboratoire Cosderma
Locations (1):
- Laboratoire COSDERMA, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No